CLINICAL TRIAL: NCT07234526
Title: Pre-Antibiotic Glucose Fluctuations and Glycemic Shock Index as a Predictor of Sepsis Severity and Clinical Outcomes in ICU Patient
Brief Title: Usage of Glucose Fluctuations as a Prognostic Marker in Septic Shock Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaban Nady Sedky Tamer, Resident physician, Assiut University
Other Study IDs: Glucose fluctuations in sepsis
Record Dates: First submitted 2025-09-17; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Glucose Fluctuations in Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine whether glucose fluctuations prior to antibiotic administration are associated with sepsis severity and poor clinical outcomes.

* To assess if the time to Glycemic Normalization after Antibiotic Initiation can be used as an Early Prognostic Indicator in Sepsis.
* To evaluate the Glycemic Shock Index (GSI) as a Combined Marker of Hemodynamic and Metabolic Stress in ICU Sepsis Patients.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition caused by the body's overwhelming response to infection. It is a major cause of death in intensive care units (ICUs) despite advances in treatment. One of the body's common responses to sepsis is a disturbance in blood sugar levels, even in patients without diabetes. These changes, known as glycemic variability, include both high and low glucose levels and rapid swings between them.

Recent studies suggest that glycemic variability the early hours of sepsis may be linked to worse outcomes, including organ failure and death .Unlike average glucose levels, these fluctuations can reflect how stressed the body is.

A newer marker called the Glycemic Shock Index (GSI) - calculated by dividing blood glucose by mean arterial pressure (MAP)- may help capture both metabolic and circulatory stress.

Another factor of interest is the time it takes for blood sugar to return to normal after starting antibiotics.

Early normalization may signal a better response to treatment, while persistent abnormal levels could predict complications.

Understanding how early glucose changes relate to sepsis severity may help us identify high-risk patients sooner. This study focuses on glucose fluctuations before antibiotics, time to glucose normalization, and GSI, and how they relate to outcomes like mortality, organ failure like AKI and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years admitted to ICU with suspected or confirmed sepsis.
* Sepsis diagnosed using Sepsis-3 criteria (infection + SOFA ≥2).
* At least 2 blood glucose readings within 6 hours prior to the first dose of antibiotics.
* at least 3 after starting antibiotics within 24 hours.

Exclusion Criteria:

* Steroid use in prior 48 hours.
* DKA, HHS, or acute pancreatitis.
* Incomplete glucose data or delayed documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care unit of assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | Baseline
  ICU mortality due to septic shock and associated glucose level fluctuations pre and post antibiotic administration
AKI | Baseline
  number of patients suffering from AKI due to septic shock

SECONDARY OUTCOMES:
Need for vasopressor support within first 24 hours. | First 24 hours of ICU admission
  Number of patients who needed norepinephrine or other vasopressors during first day of ICU admission
Length of ICU stay | Start from patient admission to ICU unti patient discharge or death for any cause (whichever comes first) up to 1 year
  Length of ICU stay until improvement or death

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abbas Al masry, Doctorate of internal medicine, Study Director

IPD SHARING:
Plan to Share IPD: Undecided
Patients may not agree